CLINICAL TRIAL: NCT03603990
Title: Effect of Vitrectomy on the Evolution of Refractory Diabetic Macular Edema: a Randomized Pragmatic Controlled Study
Brief Title: Effect of Vitrectomy on the Evolution of Refractory Diabetic Macular Edema
Acronym: VITROMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion difficulties, despite significant changes to inclusion criteria
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YLR_2018_3; 2018-A00873-52 (Other: IDRCB)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Edema; Macular Edema; Diabetic Retinopathy; Macular Degeneration; Diabetic Angiopathies; Retinal Disease
Keywords: Edema; Macular Edema; Diabetic Retinopathy; Macular Degeneration; Diabetic Angiopathies; Retinal Disease; Signs and Symptoms; Vitrectomy
MeSH Terms: conditions — Edema; Macular Edema; Diabetic Retinopathy; Macular Degeneration; Diabetic Angiopathies; Retinal Diseases; Signs and Symptoms | interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: Prospective randomized open blinded end-point (PROBE) pragmatic study
Who Masked: Outcomes Assessor
Masking Description: Although both the patient and the investigating physician will be aware of group assignment, the evaluation of the primary endpoint (visual acuity) will be performed by independent evaluators, unaware of the randomization group for each eye. The evaluation of the CSF thickness will be automatically recorded by the OCT and therefore will not be influenced by the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitrectomy (Experimental): Patient with standard pars plana vitrectomy
  During the first 6 month :Only Panretinal photocoagulation(if high-risk PDR or rubeosis iridis) may be given.
  After First Six Months : All therapies for DME may be given at the discretion of the investigator
  Interventions: Procedure: Vitrectomy
- Usual care (Active Comparator): Patients with usual care according to the investigator choice :
  During the first 6 month : All therapies for DME may be given at the discretion of the investigator during the study, except a vitrectomy.
  After First Six Months : All therapies for DME may be given at the discretion of the investigator, including a vitrectomy.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Vitrectomy — During the first 6 month :Only Panretinal photocoagulation(if high-risk PDR or rubeosis iridis) may be given.
  After First Six Months : All therapies for DME may be given at the discretion of the investigator
  Arms: Vitrectomy
Procedure: Usual care — Patients with usual care according to the investigator choice :
  During the first 6 month : All therapies for DME may be given at the discretion of the investigator during the study, except a vitrectomy.
  After First Six Months : All therapies for DME may be given at the discretion of the investigator, including a vitrectomy.
  Arms: Usual care

SUMMARY:
For patients with at least one eye with non-tractional diabetic edema refractory to 6 months of anti-VEGF injections (anti Vascular endothelial growth factor injections), a randomization is done: one group of patients will receive the standard treatment (anti-VEGF injections, switch to another anti-VEGF drug, additional photocoagulation or any other treatment except vitrectomy during the first 6 months after the randomisation) and the other group of patients will receive vitrectomy (with only additional photocoagulation during the first 6 months, then any treatment from 6 months after the randomization).

DETAILED DESCRIPTION:
In case both eyes present refractory diabetic macular edema (DME) and are eligible, the eye with the worst DME will be included and randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Type 1 or type 2 diabetes
* At least one eye with Diabetic Macular Edema (DME) (with ophthalmoscopic evidence of center-involved DME) and Failure of medical treatment considered and conducted during at least 6 months defined as follows:

  * At least 4 intravitreal anti-VEGF injections given within the prior 6 months
  * ETDRS score ≤ 78 and ≥24 (approximate Snellen equivalent 20/32 to 20/320)
  * OCT (Optical Coherence Tomography) CSF (Central Subfield) thickness value (microns): Heidelberg Spectralis: ≥305 in women; ≥320 in men
  * Less than 5 letters gain in visual acuity (VA) after the initial Anti-VEGF treatment
  * Less than 25% decrease of CMT (Central Macular Thickness) after the initial Anti-VEGF treatment
* Glated haemoglobin (HbA1c) <12 % in the last 3 months before patient inclusion

Exclusion Criteria:

* Any history of vitrectomy for the included eye
* Tractional DME: on OCT Optical Coherence Tomography), undetached posterior hyaloid membrane with anterior-posterior traction for the included eye
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110)
* Intraocular pressure ≥ 25 mmHg for the included eye
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis for the included eye
* Exam evidence of ocular toxoplasmosis for the included eye
* Aphakia for the included eye
* Ocular condition with visual acuity loss that, in the opinion of the investigator, would not improve from resolution of macular edema (e.g. foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, non-retinal condition, etc.) for the included eye
* Condition that, in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 1 month prior to enrollment
* History of macular laser photocoagulation within 3 months prior to enrollment for the included eye
* History of panretinal (scatter) photocoagulation (PRP) within 3 months prior to enrollment or anticipated need for PRP in the 6 months following enrollment into run-in phase for the included eye
* History of major ocular surgery (including scleral buckle, any intraocular surgery, etc.) within prior 3 months or anticipated within the next 6 months following enrollment for the included eye
* History of cataract extraction within 3 months prior to enrollment for the included eye
* History of prior herpetic ocular infection for the included eye
* Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to inclusion or plans to do so in the next 4 months.
* Steroid, anti-VEGF or pro-VEGF systemic treatment within 3 months prior to inclusion or anticipated use during the study
* History of chronic renal failure requiring dialysis or kidney transplant.
* Participation in an investigational trial that involved treatment with any drug that has not received regulatory approval for the indication being studied within 1 month of enrollment.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next year.
* Patient expected to move out of the area of the clinical center to an area not covered by another clinical center during the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months after randomization
  The difference between the change in the score of visual acuity between randomization and 6 months after treatment, between groups

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MER, Principal Investigator — Fondation Ophtalmologique A. de Rothschild

IPD SHARING:
Plan to Share IPD: Undecided